CLINICAL TRIAL: NCT00076180
Title: Phase I Open-Label Single-Dose Study of Humanized Mik-Beta-1 Monoclonal Antibody Directed Toward the IL-2R/IL-15R-Beta Subunit (CD122) in T Cell Large Granular Lymphocytic Leukemia
Brief Title: Hu-Mik-beta1 to Treat T-Cell Large Granular Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 040089; 04-C-0089; NCT00079196 (obsolete NCT alias)
Record Dates: First submitted 2004-01-14; First posted 2004-01-15 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01-09

CONDITIONS: T-Cell Large Granular Lymphocytic Leukemia; Leukemia, T-Cell Large Granular Lymphocytic
Keywords: cytotoxic activity against T-LGL cells; chronic lymphoproliferative disorder; T-LGL Leukemia; Natural Killer Cells; Leukemia; Lymphocytic Leukemia; T-LGL
MeSH Terms: conditions — Leukemia, Large Granular Lymphocytic; Leukemia; Leukemia, Lymphoid | interventions — Hu-Mik-beta-1 monoclonal antibody

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

ARMS (1):
- 1 (Experimental): One dose of Hu-MiK Beta-1
  Interventions: Biological: Hu-MiK-Beta-1

INTERVENTIONS:
Biological: Hu-MiK-Beta-1 — Hu-MiK-Beta-1 administered as an intravenous infusion over 90- minutes.

SUMMARY:
This study will examine the use of the humanized Mik-beta-1 (Hu-Mik-beta1) antibody in patients with T-cell large granular lymphocytic leukemia (T-LGL). Patients with T-LGL often have reduced white blood cells, red blood cells, and platelets, and increased numbers of abnormal cells called large granular lymphocytes (LGLs). Patients may have recurrent infections, anemia, or abnormal bleeding. Hu-Mik-beta1 attaches to LGL cells and blocks the action of growth factors called interleukins that stimulate LGL growth. Blocking these interleukins may stop T-LGL leukemia cells from growing. This study will determine the dose and frequency of treatment with Hu-Mik-(SqrRoot) 1 that can safely be given to patients to coat the surface of their leukemic cells with antibody, determine how long the antibody lasts in the blood after injection, and examine the side effects and possible benefits of the drug in these patients.

Patients age 18 or older with T-LGL may be eligible for this study. Candidates will be screened with a medical history and physical examination, review of pathology studies, skin biopsy, evaluation of rheumatoid arthritis if present, chest x-ray, computerized tomography (CT) scans and other imaging studies as needed, bone marrow biopsy, and blood and urine tests.

Participants will receive a single dose of Hu-Mik-beta1 by a 90-minute infusion through a vein. Groups of patients will be treated with increasing doses (0.5, 1.0, and 1.5 mg/kg) of the antibody. Patients who develop serious drug side effects are taken off the study. The treatment requires a 3- to 4-day hospital stay. In addition to Hu-Mik-(SqrRoot) 1 treatment, patients will undergo the following tests and procedures:

* Collection of blood for 8 days following the dose of Hu-Mik-beta1 to measure blood levels of the antibody.
* Follow-up visits of 1 to 2 days at 22, 29, and 43 days after the dose of the antibody and then every 3 months for a total of 9 months.
* Bone marrow aspirate and biopsy if one has not been done within 6 weeks before entering the study, and a repeat biopsy if complete remission of T-LGL is achieved after completing treatment. For the biopsy, an area of the hip is numbed and a special needle is used to draw bone marrow from the hipbone.
* Imaging studies, such as chest x-ray and CT scan of the body after completing treatment if the screening scans showed abnormalities due to the T-LGL leukemia.
* Lymph node biopsy in individuals with enlarged superficial lymph nodes due to T-LGL leukemia to see if the treatment is reaching the leukemia in the lymph nodes.

There may or may not be a direct benefit from participating in this study. However, the results may help in the treatment of future patients.

DETAILED DESCRIPTION:
Background:

* T cell large granular lymphocyte (T-LGL) leukemia is a chronic lymphoproliferative disorder associated with granulocytopenia, anemia and/or thrombocytopenia.
* Although agents such as cyclosporine and methotrexate have shown activity in T-LGL, treatment of T-LGL has remained largely undefined and symptomatic.
* The shared IL-2R/Il-15R Beta receptor (CD122) is over expressed on T-LGL cells and may stimulate growth T-LGL cells through its interaction with IL-15.
* Hu-Mik-Beta1 is a humanized monoclonal antibody that binds to IL-2R/IL-15R Beta
* Hu-Mik-Beta1 may inhibit the growth and exert cytotoxic activity against T-LGL cells.

Objectives:

* To determine the dose-limiting toxicity (DLT) and the maximum tolerated dose (MTD) of Hu-Mik-Beta1 when administered to patients with T-LGL.
* To determine the dose of Hu-Mik-Beta1 required to saturate IL-2R/IL-15R Beta (CD122) on -T-LGL cells in the peripheral blood.
* To determine the pharmacokinetics and serum die-away curve of Hu-Mik-Beta1.
* To provide preliminary information on the clinical response following single dose administration of Hu-MiK-Beta1 in patients with CD122 expressing T-LGL leukemia.

Eligibility:

--T cell large granular lymphocyte leukemia (T-LGL).

Patients must have a granulocyte count of less than 1000/microL, or hemoglobin less than 10 gm/dL, or be transfusion dependent, or platelets less than 100,000/ microL, or any combination of these unless receiving a hematopoietic growth factor.

* T-LGL cell count greater than or equal to 1000/microL (CD3 plus/CD8 plus/usually CD57 plus) by flow cytometry.
* Patients may be receiving a stable dose of a hematopoietic growth factor.

Design:

* Cohorts of 3 patients each will be treated with a single intravenous dose of Hu-Mik-Beta1 at 0.5, 1.0 or 1.5 mg/kg.
* Patients will be observed for adverse events for 6-weeks.
* Detailed pharmacokinetic studies and determination of CD122 receptor saturation will be performed.
* Response will be evaluated using hematological, flow cytometry, molecular and clinical evaluations.
* An additional 3 patients will be accrued at the highest dose or MTD to aid in design of a Phase II trial.
* Patients participating in Phase I will also be eligible to participate in Phase II.

ELIGIBILITY:
* INCLUSION CRITERIA

All patients must have histologically or cytologically confirmed T-LGL leukemia as defined by:

i. A peripheral blood smear or bone marrow biopsy/aspirate with morphological findings consistent with LGL as determined by Hematopathology section, the NIH Clinical Center, or the Laboratory of Pathology, NCI, and;

ii. An absolute C3+, CD8+, usually CD57+ cell (T-LGL) count greater than or equal to 1000/uL in the peripheral blood or bone marrow as measured by flow cytometry.

iii. At least 50% of the CD3+/CD8+ cells must also express CD122 (IL-2/15RB plus).

iv. Clonal T cell receptor (TcR) rearrangement while desirable, is not a requirement for eligibility. TcR rearrangement may be determined by Southern blotting or polymerase chain reaction (PCR).

Patients must have T-LGL-associated hemocytopenia(s)* as defined by an absolute granulocyte count (AGC) less than 1000/uL, platelet count less than100,000/uL or hemoglobin less than 9.0 gm/dL, or have required transfusion of 3 or more units of red blood cell products in the last 6 months, or any combination of these.

*Patients being treated with a stable dose of hemopoietic growth factors for greater than 4-weeks whose peripheral blood counts exceed these values are eligible for the study. A stable dose of a hematopoeitic growth factor(s) may be continued while the patient is on the study.

Patients requiring antibiotic or treatment with antiviral drugs on more than two occasions over the previous 12 months for bacterial or viral infections associated with their LGL are eligible.

Patients must be greater than or equal to 18 years of age.

Untreated patients as well as those previously treated with cyclosporine A (CsA), chemotherapy, corticosteroids, interferon, erythropoietin, IL-11, G-CSF or GM-CSF, murine MiK-Beta-1 (or having undergone splenectomy are eligible for study.

Omission of cyclosporine A, chemotherapy and interferon is required for at least 4 weeks prior to entry onto the trial. Patients on stable doses (greater than 4 weeks) of commercial erythropoietin, G-CSF, GM-CSF or IL-11 products are eligible for the study. Patients receiving corticosteroids will not be excluded. Patients receiving corticosteroids must be on a stable dose of prednisone (less than 25 mg/day) or equivalent dose steroid for at least 3 weeks before receiving MiK-B -1 on the study.

Patients must have normal renal function (serum creatinine less than or equal to 1.5 mg/dL) and hepatic function (bilirubin less than or equal to 2.0 mg/dL, SGOT, SGPT less than or equal to 2.5 fold greater than the upper limit of normal).

Patients must have a Karnofsky performance status of greater than or equal to 70%.

Patients must have a life expectancy greater than 2 months.

Patients must be able to understand and sign the Informed Consent Document.

EXCLUSION CRITERIA

Patients must have none of the following at the time of enrollment:

Symptomatic central nervous system (CNS) involvement with LGL leukemia.

Pregnant or actively nursing patients are ineligible. The effects of Hu-MiK-Beta-1 on the developing fetus and nursing infant are unknown. Female patients of childbearing potential will be tested for pregnancy within 72 hours of initiating the study.

Patients with CTC grade 4 granulocytopenia or anemia.

Patients requiring platelet transfusions in the preceding 12-months for platelet counts of less than or equal to 10,000/mm(3) or spontaneous bleeding episodes.

Patients testing positive for the human immunodeficiency virus (HIV) or human T cell lymphotrophic virus (HTLV-I/II) are ineligible, because the toxicity may be different in this population.

Patients testing positive for hepatitis B virus surface antigen (HbsAg) or antibodies to hepatitis C virus are ineligible because Hu-MiK-Beta-1 therapy might be associated with increased viral replication.

Patients receiving prior therapy with murine MiK-Beta-1 that have developed human anti-mouse (HAMA) or human anti-human (HAHA) antibodies, or that have experienced CTC grade III or greater toxicity attributable to the antibody are ineligible.

Patients with a prior history of a Grade III or greater allergic reaction related to a previously administered humanized monoclonal antibody are ineligible.

Patients with other serious concurrent medical conditions (e.g., acute myocardial infarction within 6 months, unstable angina, NYHA Class II/IV congestive heart failure, respiratory insufficiency requiring oxygen therapy, uncontrolled hypertension, symptomatic cerebrovascular disease or stroke within 6 months, receiving immunosuppression for an organ graft, etc.) that may otherwise limit their survival are not eligible.

Other malignancy within five years, unless the probability of recurrence of the prior malignancy is less than or equal to 10 percent at 5-years. Patient's curatively treated for squamous cell carcinoma and basal cell carcinoma of the skin and carcinoma in situ of the uterine cervix (CIN) or patients with a history of malignant tumor in the past that have been disease free for at least five years are also eligible for this study.

Patients with serious active infection requiring systemic anti-infective therapy.

Any physical or psychological condition that would preclude drug administration or patient compliance with the protocol or that in the opinion of the investigator may pose an additional risk in administering the study drug to the patient or that would not permit the patient to complete the study or give Informed Consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-03-01; Primary Completion 2010-11-12 (Actual); Study Completion 2019-01-09 (Actual)

PRIMARY OUTCOMES:
DLT and MTD of Hu MIK Beta 1 | 21 days
  Adverse events will be tabulated/reported by type, grade, and frequency.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Waldmann, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kohler G, Milstein C. Continuous cultures of fused cells secreting antibody of predefined specificity. Nature. 1975 Aug 7;256(5517):495-7. doi: 10.1038/256495a0. No abstract available. PMID 1172191
- [Background] Jones PT, Dear PH, Foote J, Neuberger MS, Winter G. Replacing the complementarity-determining regions in a human antibody with those from a mouse. Nature. 1986 May 29-Jun 4;321(6069):522-5. doi: 10.1038/321522a0. PMID 3713831
- [Background] Waldmann TA. Monoclonal antibodies in diagnosis and therapy. Science. 1991 Jun 21;252(5013):1657-62. doi: 10.1126/science.2047874.
- [Derived] Waldmann TA, Conlon KC, Stewart DM, Worthy TA, Janik JE, Fleisher TA, Albert PS, Figg WD, Spencer SD, Raffeld M, Decker JR, Goldman CK, Bryant BR, Petrus MN, Creekmore SP, Morris JC. Phase 1 trial of IL-15 trans presentation blockade using humanized Mikbeta1 mAb in patients with T-cell large granular lymphocytic leukemia. Blood. 2013 Jan 17;121(3):476-84. doi: 10.1182/blood-2012-08-450585. Epub 2012 Dec 3. PMID 23212516